CLINICAL TRIAL: NCT06735937
Title: The Effects of Automatic Gas-Controlled Low-Flow Anesthesia on Anesthetic Agent Consumption in Elective Surgeries: Randomized Controlled Study
Brief Title: The Effects of Automatic Gas-Controlled Low-Flow Anesthesia on Anesthetic Agent Consumption in Elective Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Elzem SEN, Assoc Prof, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019/355
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Low-flow Anesthesia
Keywords: end-tidal controlled; low flow anesthesia; consumption

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- End-tidal controlled (Experimental): Patients ventilated using end tidal controlled low-flow anesthesia
  Interventions: Other: Low flow anesthesia
- Manually controlled (Experimental): Patients ventilated using manually controlled low flow anesthesia
  Interventions: Other: Low flow anesthesia

INTERVENTIONS:
Other: Low flow anesthesia — Anesthesia management by using low flow anesthesia

SUMMARY:
In this study, we aim to compare the effects of end-tidal controlled and manually controlled low-flow anesthesia on anesthetic agent consumption in elective surgeries.

DETAILED DESCRIPTION:
In this study, we aim to compare the effects of end-tidal controlled and manually controlled low-flow anesthesia on anesthetic agent consumption in elective surgeries. This evaluation will contribute to understanding whether automated systems provide measurable advantages in clinical settings.This evaluation will contribute to understanding whether automated systems provide measurable advantages in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Aged between18-73

Exclusion Criteria:

* heart failure
* liver disease
* lung disease
* kidney disease

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
anesthesic gas consumption | At the end of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elzem Sen, Assoc Prof, Principal Investigator — University of Gaziantep
Locations (1):
- Elzem Sen, Gaziantep, Sehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No